CLINICAL TRIAL: NCT04896931
Title: New Prospective Expanded German Registry of Incidental Gallbladder Carcinoma (PERSUASION)- a Permanent Platform Including All Kind of Biliary Tract Cancers (BTC)
Status: Completed | Type: Observational
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Other Study IDs: PERSUASION
Record Dates: First submitted 2021-05-10; First posted 2021-05-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Biliary Tract Cancer; Neoadjuvant, Adjuvant and 1st Line
Keywords: biliary tract cancer; registry; molecular profiling
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — FFPE Tumor blocks, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Permanent, prospective, multicenter registry including all kind of oncological therapy lines and procedures, clinical outcome, translational research (biobanking) and QoL for all types of biliary tract cancers.

DETAILED DESCRIPTION:
Permanent, prospective, multicenter registry including all kind of oncological therapy lines and procedures, clinical outcome, translational research (biobanking) and QoL for all types of biliary tract cancers. The registry does not define any medical intervention and does not evaluate the efficacy or safety of the treatment decision made by the investigator. Every adverse event whether related to a treatment or not, will neither be documented in the trial´s eCRF nor be reported to the leading investigators of this study.

Objectives: • To establish a registry with a representative BTC-patient population in German-speaking Europe (mainly DACH region) for current and future research. The study registry is not based on a primary endpoint. The data collection includes (among basic patient-/tumor-/treatment- characteristics) the survey of quality of life (EORTC-C30), a so-called patient-reported outcome (PRO) and - if available - the collection of tissue samples for translational accompanying projects.

* Clinical data:

  * To analyse potential risk factors associated with BTC-cancer addressing clinical and biological predictors of treatment success and survival
  * To determine the course of disease and QoL throughout all applied therapy lines for patients with BTC
  * To measure progression-free, disease-free and overall survival in different BTC sub-groups, mortality and morbidity for perioperative and palliative therapy procedures
  * Recording of the therapy regimens and therapy sequences used across all treatment lines
* Molecular data (Data- and Biobanking):

  * To establish a sample collection for future molecular/genetic biomarker characterization to enable for e.g. assessment of the frequency of targetable mutations and associated therapy decisions or progression analysis in baseline and follow-up investigations

ELIGIBILITY:
Inclusion Criteria:

* Known biliary-tract cancer including intrahepatic-, extrahepatic- and gallbladder carcinomas
* age ≥18 years
* signed informed consent form
* planned for (or recently started - i.e. within the last 21 days)) neoadjuvant, adjuvant or 1st line therapy

Exclusion Criteria:

* Patients who are unable to consent because they do not understand the nature, significance and implications of the registry and therefore cannot form a rational intention
* Patient under 18 years of age
* Patient's inability to complete QoL questionnaire or answer the questions.
* Second-line or further palliative therapies if the patient's first-line therapy was not documented within the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Permanent, prospective, multicenter registry including all kind of oncological therapy lines and procedures, clinical outcome, translational research (biobanking) and QoL for all types of biliary tract cancers.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Establishment of BTC population | Through study completion, an average of 2 years
  To establish a representative BTC-patient population in German-speaking Europe in an agile platform study design for future research

SECONDARY OUTCOMES:
analyse potential risk factors associated with BTC-cancer | Through study completion, an average of 2 years
  Correlate medical history with patient outcome, find prevalent medical history associated with BTC chancer
The course of Quality of Life (QoL) throughout the entire course of therapy for patients with BTC | Through study completion, an average of 2 years
  EORTC-QLQC30 according to EORTC scoring manual
PFS | Through study completion, an average of 2 years
  progression-free survival in different BTC subgroups and therapy lines. As for the main objective, there is no formal secondary endpoint in a registry study. Therfore, in this section we will explain the main data to be collected and the main outcome measures.
DFS | Through study completion, an average of 2 years
  disease-free survival in different BTC subgroups and therapy lines. As for the main objective, there is no formal secondary endpoint in a registry study. Therfore, in this section we will explain the main data to be collected and the main outcome measures.
OS | Through study completion, an average of 2 years
  overall survival in different BTC subgroups and therapy lines. As for the main objective, there is no formal secondary endpoint in a registry study. Therfore, in this section we will explain the main data to be collected and the main outcome measures.
mortality | Through study completion, an average of 2 years
  mortality for perioperative and palliative therapy procedures
morbidity | Through study completion, an average of 2 years
  morbidity for perioperative and palliative therapy procedures
establishment of sample collection (tumorblocks and blood) | Through study completion, an average of 2 years
  establish a sample collection for future molecular/genetic biomarker characterization

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Götze, PD Dr., Study Director — Krankenhaus Nordwest GmbH
Locations (25):
- Germany (25):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Medius Klinik Ostfildern-Ruit, Ostfildern, Baden-Wurttemberg
  - Klinikum St. Marien Amberg, Amberg, Bavaria
  - Helios Amper-Klinikum Dachau, Dachau, Bavaria
  - Donau-Isar-Klinikum Deggendorf, Deggendorf, Bavaria
  - ÜBAG-Medizinisches Versorgungszentrum. Dr. Vehling-Kaiser GmbH, Landshut, Bavaria
  - LMU Klinikum Campus Großhadern, München, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - HELIOS Klinikum Bad Saarow, Bad Saarow, Brandenburg
  - Ambulantes Zentrum für Hämatologie und Onkologie, Cottbus, Brandenburg
  - Universitätsklinikum Gießen, Giessen, Hesse
  - St. Bernward Krankenhaus Hildesheim, Hildesheim, Lower Saxony
  - Klinikum Oldenburg, Oldenburg, Lower Saxony
  - Klinikum Südstadt Rostock, Rostock, Mecklenburg-Vorpommern
  - Krankenhaus Maria-Hilf Krefeld, Krefeld, North Rhine-Westphalia
  - Klinikum Lippe Lemgo, Lemgo, North Rhine-Westphalia
  - Onkologische Schwerpunktpraxis Speyer, Speyer, Rhineland-Palatinate
  - Onkozentrum Dresden, Dresden, Saxony
  - Onkologische Schwerpunktpraxis Freital, Freital, Saxony
  - Universitäres Krebszentrum Universitätsklinikum Leipzig (UCCL), Leipzig, Saxony
  - Onkologische Schwerpunktpraxis, Naunhof, Saxony
  - Elblandklinikum Riesa, Riesa, Saxony
  - Gemeinschaftspraxis für Onkologie und Hämatologie, Erfurt, Thuringia
  - Charité - Universitätsmedizin Berlin, Berlin
  - Krankenhaus Nordwest GmbH, Frankfurt

IPD SHARING:
Plan to Share IPD: No